CLINICAL TRIAL: NCT01812278
Title: Randomized Trial of Web-Delivered Acceptance Therapy for Smoking Cessation
Brief Title: Randomized Trial of Web-Delivered Acceptance Therapy for Smoking Cessation (WebQuit)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Kaiser Permanente (Other); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7859; NCI-2019-06975 (Registry Identifier: NCI / CTRP); R01CA166646 (NIH)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2019-12

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Acceptance and Commitment Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT (Experimental): Acceptance & Commitment Therapy
  Interventions: Behavioral: ACT
- CBT (Active Comparator): Cognitive Behavioral Therapy
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: ACT
  Other Names: Acceptance & Commitment Therapy
  Arms: ACT
Behavioral: CBT
  Other Names: Cognitive Behavioral Therapy
  Arms: CBT

SUMMARY:
The goal of this study is to determine whether the ACT website provides higher quit rates than a current standard smoking cessation website.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* smokes at least five cigarettes daily for at least past 12 months
* wants to quit in next 30 days
* willing to be randomly assigned to either group
* resides in US
* has at least weekly access to a high speed Internet connection and email
* willing and able to read in English
* not participating in other smoking cessation interventions (including our other intervention studies
* has never used the Smokefree.gov website
* willing to complete all three follow-up surveys
* provide email, phone, and mailing address
* provide contact information for two collaterals (e.g., relatives).
* does not have family, friends, or other household members participating

Exclusion Criteria:

* The exclusion criteria are the opposite of the inclusion criteria above.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2637 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
30-day point prevalence abstinence | 12 month post randomization
  No smoking in the past 30 days, as reported 12 month post treatment.

SECONDARY OUTCOMES:
7-day, 24-hour, and 30-day point prevalence quit rates | 3 months, 6 months, and 12 months post treatment
  12 months: 24-hour and 7-day point prevalence quit rates. 3 and 6 months: 24-hour, 7-day, and 30-day point prevalence quit rates. Across 3, 6, and 12 month timepoints, the repeated 30-day point prevalence abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bricker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Santiago-Torres M, Kwon DM, Mull KE, Sullivan BM, Ahluwalia JS, Alexander AC, Nollen NL, Bricker JB. Efficacy of Web-Delivered Acceptance and Commitment Therapy (ACT) for Helping Black Adults Quit Smoking. J Racial Ethn Health Disparities. 2023 Dec;10(6):2816-2825. doi: 10.1007/s40615-022-01458-5. Epub 2022 Nov 21. PMID 36414931
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700
- [Derived] Watson NL, Heffner JL, Mull KE, McClure JB, Bricker JB. Comparing Treatment Acceptability and 12-Month Cessation Rates in Response to Web-Based Smoking Interventions Among Smokers Who Do and Do Not Screen Positive for Affective Disorders: Secondary Analysis. J Med Internet Res. 2019 Jun 19;21(6):e13500. doi: 10.2196/13500. PMID 31219052
- [Derived] Watson NL, Mull KE, Heffner JL, McClure JB, Bricker JB. Participant Recruitment and Retention in Remote eHealth Intervention Trials: Methods and Lessons Learned From a Large Randomized Controlled Trial of Two Web-Based Smoking Interventions. J Med Internet Res. 2018 Aug 24;20(8):e10351. doi: 10.2196/10351. PMID 30143479
- [Derived] Bricker JB, Sridharan V, Zhu Y, Mull KE, Heffner JL, Watson NL, McClure JB, Di C. Trajectories of 12-Month Usage Patterns for Two Smoking Cessation Websites: Exploring How Users Engage Over Time. J Med Internet Res. 2018 Apr 20;20(4):e10143. doi: 10.2196/10143. PMID 29678799